CLINICAL TRIAL: NCT06840522
Title: The Importance of Tailored Education And Device Handling for Asthmatic Patients
Acronym: TEACH
Status: Not yet recruiting | Type: Observational
Sponsor: Chiesi Hungary Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DE-HI/2024/01
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: Inhalation treatment; Lung deposition
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma patients on GINA steps 3 and 4 receiving Foster Nexthaler treatment: Asthma patients above the age of 18 years. Uncontrolled according to the physician's clinical assessment despite the use of appropriate therapy of Step 2 or 3, according to GINA guidelines. Patients who are eligible for the use of Foster Nexthaler 100/6 mcg according to the SmPC. Inhaled asthma therapy was changed independent from the study to Foster Nexthaler 100/6 mcg DPI maximum 1 week prior to OR on the day of study inclusion. Spirometry was performed as part of routine clinical practice
  . Patient able to use their Foster Nexthaler device properly after education on inhaler technique. Patient provided written, informed consent to study participation

SUMMARY:
Significant advancements have been made in asthma medication over the past decades. Highly effective treatments are available for patients; however, both adherence and proper device usage remain below the desired levels, based on our experience and literature data. Despite the availability of numerous excellent drug-device combinations, personalized treatment for patients is still not adequately addressed.

In the present study, the aim is to improve patient compliance and educate symptomatic, partially, or uncontrolled asthma patients on the correct use of a specific inhalation device (Nexthaler). Considering the characteristics of the medication, the patient's lung function data, inhalation technique, and drug retention time can help estimate the expected lung deposition of the medication. By refining the inhalation technique under the guidance of the treating physician, it is hypothesized that the expected therapeutic effects of the medication may improve.

DETAILED DESCRIPTION:
Eligible Patient Population:

Patients on GINA step 2-4 therapy who are partially or uncontrolled (ACT <25) and are receiving Foster Nexthaler® therapy as per prescribing guidelines, regardless of the study. Patients on GINA step 3 therapy receive a low-dose ICS-formoterol regimen (2x1 inhalations of Foster Nexthaler® 100/6 μg), while those on GINA step 4 receive a medium-dose ICS-formoterol regimen (2x2 inhalations of Foster Nexthaler® 100/6 μg). Whenever possible, Foster Nexthaler® 100/6 μg is used as a reliever medication following the MART principles. If the treating physician opts for salbutamol (Ventolin®, Buventol®) instead, the patient may still be included in the study, provided justification is given, considering the difficulty of training with multiple inhalation devices (pMDI and DPI with different characteristics).

Study Procedures:

Lung function tests will be performed on enrolled patients. The investigating physician will evaluate the recorded spirometry curves, which will be used for computer modeling to assess pulmonary drug deposition. The spirometry curves are also useful for evaluating the patient's condition and monitoring progress.

During the study visits (V1 - enrollment, V2 - 1 month, V3 - 3 months), the following data will be recorded: patient demographics, medical history, treatment details, risk factors, medication adherence (based on prescription refills and patient self-report), and quality of life assessment. Data collection, particularly questionnaire results, will follow the daily routine of the study center.

Study Objective:

The aim is to demonstrate that patient education on using a specific inhalation device (Foster Nexthaler®), optimizing inhalation technique (prolonging breath-hold time), and the resulting increased drug deposition lead to measurable clinical benefits, improved asthma control, and higher ACT scores.

Education on inhaler use and practicing optimal inhalation techniques are expected to improve lung function, maintain adherence, and reduce the need for rescue medication.

ELIGIBILITY:
Inclusion Criteria:

1. Physician-confirmed clinical diagnosis of asthma according to GINA guidelines
2. Uncontrolled asthma according to the physician's clinical assessment despite the use of appropriate therapy of Step 2 or 3, according to GINA guidelines
3. Patients who are eligible for the use of Foster Nexthaler 100/6 mcg according to the SmPC
4. Inhaled asthma therapy was changed independent from the study to Foster Nexthaler 100/6 mcg DPI maximum 1 week prior to OR on the day of study inclusion
5. Spirometry was performed as part of routine clinical practice
6. Patient able to use their Foster Nexthaler device properly after education on inhaler technique
7. Patient provided written, informed consent to study participation
8. Patient ≥ 18 years of age

Exclusion Criteria:

1. Participation in any clinical trial, 30 days prior to inclusion
2. Patient is unable to execute a spirometry test
3. Patients hospitalized due to an exacerbation of their asthma within the last 4 weeks prior to enrolment.
4. Patients with other significant diseases of the respiratory system or other organ systems that may significantly contribute to asthma symptoms (such as severe heart failure, symptomatic anaemia, functional respiratory disorders, malignant diseases etc.) according to the physician's clinical assessment.
5. Continuous use of oral corticosteroids (>5 mg prednisolone/day or >4 mg methylprednisolone/day)
6. Use of continuous oxygen therapy
7. Use of biologics for asthma treatment
8. All exclusion criteria listed in Foster Nexthaler 100/6 SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients, treated in routine clinical practice, symptomatic on previous therapy, and switched to Foster 100/6 micrograms in Nexthaler device, irrespective of study inclusion,
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary deposition | 3 months
  Difference of pulmonary deposition between patients performing different lengths of breath hold and it's changes after 3 months of treatment.
Asthma control questionnaire | 3 months
  Change in asthma control questionnaire (ACQ-6) scores after 3 months of treatment between patients performing different lengths of breath hold.

SECONDARY OUTCOMES:
Asthma control | 3 months
  Proportion of patients achieving improvement in asthma control at Visit 3 between patients performing different lengths of breath hold
Lung function | 3 months
  Change in spirometry parameters: Forced expiratory volume in 1 second, Forced vital capacity and their ratio, at Visit 3, compared to the baseline between patients performing different lengths of breath hold
Rescue medication | 3 months
  Change in the need for rescue medications at Visit 3, compared to the baseline between patients performing different lengths of breath hold
Adherence | 3 months
  Changes in treatment adherence based on prescription filled at Visit 3, compared to the baseline between patients performing different lengths of breath hold
Fractional exhaled nitric oxide | 3 months
  Change in fractional exhaled nitric oxide (FeNO) values at Visit 3 (count and percentage of patients with FeNO above 20 ppb) between patients performing different lengths of breath hold
Health related quality of life | 3 months
  To assess changes in quality of life in EQ-5D-5L domains after 3 months of treatment compared to baseline. Scale on a level of five
Adherence self report | 3 months
  To assess changes itest of adherence to inhalers questionnaire (TAI-12) after 3 months of treatment compared to baseline.

CONTACTS AND LOCATIONS:
Locations (6):
- Hungary (6):
  - National Korányi Institute of Pulmonology, Budapest
  - Department of Pulmonology and Allergology, Csornai MArgit Hospital, Csorna
  - Department of Pulmonology, Debrecen University, Debrecen
  - Pulmonology Outpatient Clinic of Dunakeszi, Dunakeszi
  - Department of Pulmonology, University of Szeged, Szeged
  - Calvinist Pulmonology Centre, Törökbálint

IPD SHARING:
Plan to Share IPD: No